CLINICAL TRIAL: NCT02365831
Title: Evaluation of Medical Treatments in MBC HER2 Negative Patients in Italy - Observational Study
Brief Title: Observation of Medical Treatments in MBC HER2-negative Patients
Acronym: AMBRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Consorzio Oncotech (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: GIM13-AMBRA
Record Dates: First submitted 2014-12-15; First posted 2015-02-19 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Metastatic Breast Cancer
Keywords: MBC; breast; metastatic; cancer; HER2
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Histologic samples for the evaluation of metastatic breast cancer according to biological subtype definition (Luminal A, Luminal B, HER2 positive, triple-negative).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prospective: Observation of treatment management of patients with metastatic breast cancer that have been treated or not with hormonal therapy and candidate for a first line chemotherapeutic treatment in the years 2014-2015 will be observed until the end of the study.
  Interventions: Other: Observation of treatment management
- Retrospective: Observation of treatment management of patients with metastatic breast cancer that have been treated with a first, second or following line of chemotherapeutic treatment for metastatic disease in the years 2012-2013.
  Interventions: Other: Observation of treatment management

INTERVENTIONS:
Other: Observation of treatment management — Group/cohort

SUMMARY:
While therapeutic strategies for HER2-positive breast cancer are well defined, there is not a standard strategy for HER2-negative tumors.

Because of lack of information related to the the factors affecting the choice of a particular treatment strategy, as well as the optimization of the correct sequence of treatments, the choice of the treatment for the advanced disease remains highly empirical and may differ significantly among the different cancer centers.

The purpose of this study is the observation of a cohort of patients with metastatic HER2-negative in terms of:

1. the choice of chemotherapy treatments starting from the first line of treatment;
2. factors that may influence these choices;
3. correlation among the characteristics of patients (age, menopausal status, etc.) and type of adjuvant and metastatic treatment ;
4. clinical outcome (pattern of relapse, time from diagnosis, etc.);
5. evaluation of the adherence to the literature's recommendations for therapeutic sequences in clinical practice.

DETAILED DESCRIPTION:
In particular, the attention will be on those factors, largely discussed in the literature, that predominantly guide the choice among different therapeutic approaches such as:

* metastatic sites;
* hormone receptor status;
* disease-free interval;
* grading;
* response to a previous treatment with hormonal therapy or chemotherapy. The primary objective is the description of medical therapeutic strategies for the first, the second and the subsequent lines of chemotherapy in a cohort of patients with HER2-negative metastatic breast cancer and the evaluation of the possible correlation between the choice of treatment, in the adjuvant phase or for the metastatic disease and also for the patients' characteristics (age, menopausal status, comorbidity).

the secondary objectives are:

* Analyze the "Time to Treatment Change", defined as the interval of time that elapses from the start of chemotherapy to the discontinuation or the occurrence of any other event. This finding is of a particular clinical relevance, since randomized trials using the "Time To Progression" (TTP) as a measure of effectiveness of the treatment in the study, but this time parameter may not correspond to what is observed in clinical practice, where the revaluations of disease are not conducted at preset intervals as is in the case of controlled clinical trials.
* Evaluate the correlation between the characteristics of the patients and the choice of the type of chemotherapy.
* Assess the potential correlation between the type of adjuvant therapy and the type of response obtained with the first-line treatment and between the answer to this last therapy line and second/third one.
* Assess the adherence to the literature's recommendations (Consensus Conferences and Guide-lines) of the choices between the sequential therapy vs the combination therapy in different lines of treatment (first, second, third line) of the metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HER2-negative metastatic breast cancer (Stage IV), that have received or not the endocrine therapy for the metastatic disease and that are candidate for the first-line chemotherapy treatment in the years 2014-2015 (prospective cohort), or patients that have received a treatment of first, second or subsequent-line of chemotherapy for the metastatic disease in the years 2012-2013 (retrospective cohort).
2. Age > 18 years
3. Availability of all information required by the study, in particular:

   * histology
   * hormone receptor status
   * grading
   * stage of disease at diagnosis
   * type of surgery for the primary tumor
   * type of adjuvant therapy (chemotherapy or hormone therapy)
   * type of medication received as adjuvant therapy
   * date and seat of the relapse
   * type of treatment received for the first / second / third-line of treatment of metastatic disease (chemotherapy or hormone therapy)
   * type of chemotherapy regimen used and details about the medication, date and seat of disease progression
4. Written informed consent (in case of the impossibility to obtain the consent in writing, eg, death of the patient, the data will be collected as required by the Guarantor, OJ N.72 of March 26, 2012)

Exclusion Criteria:

1. Patients with metastatic disease at diagnosis
2. Patients with HER2-positive breast
3. Participation in clinical research protocols, both for the retrospective cohort and for the perspective one

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients from Italy with metastatic breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number subsequent lines of treatment. | Outcome 1 assessed up to 24 months (2012 until 2016 where applicable)
  Evaluation of correlation between treatment choice and patient characteristic ( age, menopausal status, comorbidity).

SECONDARY OUTCOMES:
Time to Treatment Change | Outcome 2 assessed up to 24 months (2012 until 2016 where applicable)
  evaluation of the time interval between the begin of chemotherapic treatment and its interruption.
Correlation between the type of adjuvant therapy and the type of response to the treatment | Outcome 3 assessed up to 24 months (2012 until 2016 where applicable)
Evaluation of the adherence to the Consensus Conferences and Guidelines concerning the choice between the sequential therapies versus the combination therapies ( first, second, third line) | Outcome 4 assessed up to 24 months (2012 until 2016 where applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Cazzaniga, MD, Principal Investigator — Azienda Ospedaliera San Gerardo-Oncologia Medica (Saint Gerard Hospital-Medical Oncology)
Locations (1):
- A.O. San Gerardo, Monza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez EA, Suman VJ, Davidson NE, Gralow JR, Kaufman PA, Visscher DW, Chen B, Ingle JN, Dakhil SR, Zujewski J, Moreno-Aspitia A, Pisansky TM, Jenkins RB. Sequential versus concurrent trastuzumab in adjuvant chemotherapy for breast cancer. J Clin Oncol. 2011 Dec 1;29(34):4491-7. doi: 10.1200/JCO.2011.36.7045. Epub 2011 Oct 31. PMID 22042958
- [Background] Cazzaniga ME, Mustacchi G, Pronzato P, De Matteis A, Di Costanzo F, Floriani I; NORA Study Group. Adjuvant systemic treatment of early breast cancer: the NORA study. Ann Oncol. 2006 Sep;17(9):1386-92. doi: 10.1093/annonc/mdl132. Epub 2006 Jun 21. PMID 16790520
- [Background] Smith I, Procter M, Gelber RD, Guillaume S, Feyereislova A, Dowsett M, Goldhirsch A, Untch M, Mariani G, Baselga J, Kaufmann M, Cameron D, Bell R, Bergh J, Coleman R, Wardley A, Harbeck N, Lopez RI, Mallmann P, Gelmon K, Wilcken N, Wist E, Sanchez Rovira P, Piccart-Gebhart MJ; HERA study team. 2-year follow-up of trastuzumab after adjuvant chemotherapy in HER2-positive breast cancer: a randomised controlled trial. Lancet. 2007 Jan 6;369(9555):29-36. doi: 10.1016/S0140-6736(07)60028-2. PMID 17208639
- [Result] O'Shaughnessy JA, Brufsky AM. RiBBON 1 and RiBBON 2: phase III trials of bevacizumab with standard chemotherapy for metastatic breast cancer. Clin Breast Cancer. 2008 Aug;8(4):370-3. doi: 10.3816/CBC.2008.n.045. No abstract available. PMID 18757267
- [Result] Slamon D, Eiermann W, Robert N, Pienkowski T, Martin M, Press M, Mackey J, Glaspy J, Chan A, Pawlicki M, Pinter T, Valero V, Liu MC, Sauter G, von Minckwitz G, Visco F, Bee V, Buyse M, Bendahmane B, Tabah-Fisch I, Lindsay MA, Riva A, Crown J; Breast Cancer International Research Group. Adjuvant trastuzumab in HER2-positive breast cancer. N Engl J Med. 2011 Oct 6;365(14):1273-83. doi: 10.1056/NEJMoa0910383. PMID 21991949
- [Result] Piccart-Gebhart MJ, Procter M, Leyland-Jones B, Goldhirsch A, Untch M, Smith I, Gianni L, Baselga J, Bell R, Jackisch C, Cameron D, Dowsett M, Barrios CH, Steger G, Huang CS, Andersson M, Inbar M, Lichinitser M, Lang I, Nitz U, Iwata H, Thomssen C, Lohrisch C, Suter TM, Ruschoff J, Suto T, Greatorex V, Ward C, Straehle C, McFadden E, Dolci MS, Gelber RD; Herceptin Adjuvant (HERA) Trial Study Team. Trastuzumab after adjuvant chemotherapy in HER2-positive breast cancer. N Engl J Med. 2005 Oct 20;353(16):1659-72. doi: 10.1056/NEJMoa052306. PMID 16236737
- [Result] Gianni L, Dafni U, Gelber RD, Azambuja E, Muehlbauer S, Goldhirsch A, Untch M, Smith I, Baselga J, Jackisch C, Cameron D, Mano M, Pedrini JL, Veronesi A, Mendiola C, Pluzanska A, Semiglazov V, Vrdoljak E, Eckart MJ, Shen Z, Skiadopoulos G, Procter M, Pritchard KI, Piccart-Gebhart MJ, Bell R; Herceptin Adjuvant (HERA) Trial Study Team. Treatment with trastuzumab for 1 year after adjuvant chemotherapy in patients with HER2-positive early breast cancer: a 4-year follow-up of a randomised controlled trial. Lancet Oncol. 2011 Mar;12(3):236-44. doi: 10.1016/S1470-2045(11)70033-X. Epub 2011 Feb 25. PMID 21354370
- [Result] Clavarezza M, Mustacchi G, Casadei Gardini A, Del Mastro L, De Matteis A, Riccardi F, Adamo V, Aitini E, Amoroso D, Marchetti P, Gori S, Carrozza F, Maiello E, Giotta F, Dondi D, Venturini M. Biological characterization and selection criteria of adjuvant chemotherapy for early breast cancer: experience from the Italian observational NEMESI study. BMC Cancer. 2012 Jun 6;12:216. doi: 10.1186/1471-2407-12-216. PMID 22672524
- [Result] Gennari A, Stockler M, Puntoni M, Sormani M, Nanni O, Amadori D, Wilcken N, D'Amico M, DeCensi A, Bruzzi P. Duration of chemotherapy for metastatic breast cancer: a systematic review and meta-analysis of randomized clinical trials. J Clin Oncol. 2011 Jun 1;29(16):2144-9. doi: 10.1200/JCO.2010.31.5374. Epub 2011 Apr 4. PMID 21464403
- [Result] Kennecke H, Yerushalmi R, Woods R, Cheang MC, Voduc D, Speers CH, Nielsen TO, Gelmon K. Metastatic behavior of breast cancer subtypes. J Clin Oncol. 2010 Jul 10;28(20):3271-7. doi: 10.1200/JCO.2009.25.9820. Epub 2010 May 24. PMID 20498394
- [Result] Arvold ND, Taghian AG, Niemierko A, Abi Raad RF, Sreedhara M, Nguyen PL, Bellon JR, Wong JS, Smith BL, Harris JR. Age, breast cancer subtype approximation, and local recurrence after breast-conserving therapy. J Clin Oncol. 2011 Oct 10;29(29):3885-91. doi: 10.1200/JCO.2011.36.1105. Epub 2011 Sep 6. PMID 21900114
- [Result] Beslija S, Bonneterre J, Burstein HJ, Cocquyt V, Gnant M, Heinemann V, Jassem J, Kostler WJ, Krainer M, Menard S, Petit T, Petruzelka L, Possinger K, Schmid P, Stadtmauer E, Stockler M, Van Belle S, Vogel C, Wilcken N, Wiltschke C, Zielinski CC, Zwierzina H; Central European Cooperative Oncology Group (CECOG). Third consensus on medical treatment of metastatic breast cancer. Ann Oncol. 2009 Nov;20(11):1771-85. doi: 10.1093/annonc/mdp261. Epub 2009 Jul 16. PMID 19608616
- [Result] Cazzaniga M, Pronzato P, Leto di Priolo SL, De Matteis A, Di Costanzo F, Passalacqua R, Rosso R, Torri V. Patterns of relapse and modalities of treatment of breast cancer: the 'IRIS' Project, a multicenter observational study. Oncology. 2004;66(4):260-8. doi: 10.1159/000078325. PMID 15218292
- [Result] Newcombe RG. Two-sided confidence intervals for the single proportion: comparison of seven methods. Stat Med. 1998 Apr 30;17(8):857-72. doi: 10.1002/(sici)1097-0258(19980430)17:83.0.co;2-e. PMID 9595616